CLINICAL TRIAL: NCT00799383
Title: Counteracting Risperidone-Induced Hyperprolactinemia in Youths
Brief Title: Calcium and Vitamin D to Optimize Bone Mass in Boys With Risperidone-induced Hyperprolactinemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chadi A. Calarge (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Children's Miracle Network (Other)
Responsible Party: Sponsor-Investigator, Chadi A. Calarge, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200807730; K23MH085005 (NIH)
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Risperidone-induced Hyperprolactinemia
Keywords: Risperidone; hyperprolactinemia; children; adolescents; antipsychotics; prevention; calcium; vitamin D; Risperidone-induced hyperprolactinemia
MeSH Terms: conditions — Hyperprolactinemia | interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Calcium and Vitamin D (Experimental): Calcium carbonate 625mg and vitamin D 200IU will be administered, orally, twice a day for a nine-month period.
  Interventions: Drug: Calcium and Vitamin D
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Calcium and Vitamin D — Calcium carbonate 625mg and vitamin D 200IU will be administered, orally, twice a day for a nine-month period.
  Other Names: Ca+VitD
  Arms: Calcium and Vitamin D
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether calcium and vitamin D supplementation, over a nine-month period, optimizes bone mineralization in boys with risperidone-induced hyperprolactinemia. We hypothesize that, by the end of the stuy, children in the supplementation group will have higher bone mineral density compared to those in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Males (age range: 5-17yo; inclusive), in treatment with risperidone for ≥ one year.
2. The participants must have two measurements of prolactin ≥ 18.4 ng/ml, obtained within a week.
3. IQ > 35-40 (≥ Moderate intellectual disability).
4. An adult parent/guardian must be available to provide consent and dispense study medication.

Exclusion Criteria:

1. Chronic disorders involving a vital organ (heart, lung, liver, kidney, brain), metabolic diseases (e.g., diabetes, hypo- or hyperparathyroidism, hypo- or hyperthyroidism, growth hormone deficiency), other skeletal diseases (e.g., Paget's disease, osteogenesis imperfecta, rheumatoid arthritis), chronic use of drugs affecting bone metabolism (e.g., corticosteroids), and malnutrition conditions (e.g., chronic diarrhea, inflammatory bowel disease), congenital disorders, or lead poisoning.
2. Participants receiving calcium or multivitamins in the previous three months.
3. A history of renal calculi and fasting random urine calcium/creatinine ratio > 0.2 or any other medical disorder that contraindicates the use of calcium or vitamin D (e.g., hypercalcemic states, hypercoagulability disorders, vitamin D toxicity, malabsorption syndrome, or hypersensitivity to vitamin D products).
4. Laboratory values outside the normal range, except for prolactin, unless the deviations were not clinically significant (e.g. TSH < 10 μIU/ml (76)).
5. Inability to cooperate with the BMD measurements.
6. Bilateral wrist or forearm fractures.
7. Eating disorders.
8. Non-compliance with the prescribed psychiatric treatment as reflected by an undetectable combined risperidone and 9-hydroxy risperidone blood concentration.
9. Plans to move out of State within the next 9 months.

Ages: 5 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2008-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Calarge, M.D., Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Calarge CA, Mills JA, Ziegler EE, Schlechte JA. Calcium and Vitamin D Supplementation in Boys with Risperidone-Induced Hyperprolactinemia: A Randomized, Placebo-Controlled Pilot Study. J Child Adolesc Psychopharmacol. 2018 Mar;28(2):145-150. doi: 10.1089/cap.2017.0104. Epub 2017 Nov 7. PMID 29112461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 02/2009 and 11/2013, medically-healthy 5 to 17 year-old risperidone-treated boys were enrolled, via screening of the electronic medical records, referrals, and word of mouth.
Pre-assignment Details: Participants were required to have been in treatment with risperidone for at least one year.
  They should have had a prolactin concentration ≥ 18.4 ng/ml on two occasions, within one week.
Groups:
- Calcium+VitD: Calcium and Vitamin D: Calcium carbonate 625mg and vitamin D 200IU will be administered, orally, twice a day for a nine-month period.
- Placebo: Placebo administered in similarly looking capsules.
Period: Overall Study
Arm/Group | Calcium+VitD | Placebo
Started | 23 | 24
Completed | 20 | 18
Not Completed | 3 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Urinary Calcium/Creatinine > 0.2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Calcium+VitD; Placebo: Calcium and Vitamin D: Calcium carbonate 625mg and vitamin D 200IU will be administered, orally, twice a day for a nine-month period.
  I labelled the intervention type as "drug", even though "dietary supplement" would be more appropriate as the system sent the following error message:
  ERROR: An IND/IDE study must have at least one intervention of type: Drug, Device, Biological/Vaccine, Radiation or Genetic.
- Total: Total of all reporting groups
Arm/Group | Calcium+VitD | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.0) | 12.1 (3.0) | 11.5 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 23 | 24 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 21 | 24 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Total Body Less Head Bone Mineral Content Z-score [Mean (Standard Deviation); unit: Z-score] — This measure is based on a whole-body dual energy x-ray absorptiometry (DXA) scan.
  Z-score | 0.10 (0.79) | 0.12 (0.68) | 0.11 (0.73)
Trabecular Bone Mineral Density, mg/cm3 [Mean (Standard Deviation); unit: mg/cm3] — Population: The number at baseline is smaller than the randomized number because bone scans with movement artifact were discarded
  mg/cm3
    number analyzed (Participants) | 22 | 21 | 43
    (all) | 192.9 (31.1) | 197.2 (43.9) | 195.0 (37.5)

OUTCOME MEASURES:

1. Primary Outcome: Trabecular Bone Mineral Density in the Ultradistal Radius
Description: Peripheral quantitative computed tomography (pQCT) scan was obtained at the 4% and 20% sites of the nondominant radius to estimate trabecular and cortical BMD, respectively. A Stratec XCT-2000 scanner, software version 6.0 (Stratec, Inc., Pforzheim, Germany),was used. Trabecular BMD was measured as the mean density of the 85% central area of the bone's cross-section.
  Outcomes were measured at baseline, 18 weeks, and 36 weeks later.
Time Frame: 36 weeks
Population: The number at baseline is smaller than the randomized number because bone scans with movement artifact were discarded. At late time points, the sample size reflects both attrition and exclusion due to movement artifact.
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 22 | 21
mg/cm^3
  Baseline | 192.9 (31.1) | 197.2 (43.9)
  At 18 Weeks: number analyzed (Participants) | 20 | 16
  At 18 Weeks | 191.0 (38.4) | 194.6 (41.2)
  At 36 Weeks: number analyzed (Participants) | 19 | 12
  At 36 Weeks | 195.7 (36.9) | 213.1 (42.1)

2. Primary Outcome: Total Body Bone Mineral Content
Description: Outcomes were measured at baseline, 18 weeks, and 36 weeks later.
Time Frame: 36 weeks
Population: Numbers below reflect attrition.
Measure: Mean (Standard Deviation); unit: Z score (age-sex-height-race specific)
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 23 | 24
Z score (age-sex-height-race specific)
  At Baseline | 0.10 (0.79) | 0.12 (0.68)
  At 18 Weeks: number analyzed (Participants) | 20 | 19
  At 18 Weeks | 0.24 (0.81) | 0.23 (0.76)
  At 36 Weeks: number analyzed (Participants) | 20 | 18
  At 36 Weeks | 0.20 (0.86) | 0.17 (0.78)

3. Secondary Outcome: Bone Strength Index, mg2/mm4
Description: Measured at the 4% radius site.
Time Frame: 36 weeks
Population: Sample size is smaller because scans with movement artifact were removed at baseline. At follow up, attrition also contributed.
Measure: Mean (Standard Deviation); unit: mg^2/mm^4
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 22 | 21
mg^2/mm^4
  Baseline | 19.8 (8.1) | 25.3 (15.9)
  week 18: number analyzed (Participants) | 20 | 16
  week 18 | 21.0 (9.1) | 22.9 (14.3)
  week 36: number analyzed (Participants) | 19 | 12
  week 36 | 23.1 (9.6) | 26.1 (14.5)

4. Secondary Outcome: Cortical Bone Mineral Density
Description: This was measured at the 20% radius site.
Time Frame: 36 weeks
Population: Sample size reduced due to exclusion of scans with movement artifact and, in later visits, due to attrition as well.
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 18 | 20
mg/cm^3
  Baseline | 1059.6 (34.8) | 1063.2 (30.6)
  week 18: number analyzed (Participants) | 18 | 16
  week 18 | 1062.8 (34.5) | 1060.2 (27.1)
  week 36: number analyzed (Participants) | 16 | 20
  week 36 | 1069.3 (31.8) | 1058.7 (27.4)

5. Secondary Outcome: Cortical Thickness
Description: This was measured at the 20% radius site.
Time Frame: 36 weeks
Population: Sample size reduced due to exclusion of scans with movement artifact and, in later visits, due to attrition as well.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 18 | 20
mm
  Baseline | 2.25 (0.32) | 2.34 (0.50)
  week 18: number analyzed (Participants) | 18 | 16
  week 18 | 2.25 (0.34) | 2.26 (0.45)
  week 36: number analyzed (Participants) | 16 | 16
  week 36 | 2.32 (0.35) | 2.34 (0.44)

6. Secondary Outcome: Periosteal Circumference
Description: This was measured at the 20% radius site.
Time Frame: 36 weeks
Population: Sample size reduced due to exclusion of scans with movement artifact and, in later visits, due to attrition as well.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 18 | 20
mm
  Baseline | 30.1 (4.3) | 32.4 (5.4)
  week 18: number analyzed (Participants) | 18 | 16
  week 18 | 31.2 (4.3) | 32.6 (6.1)
  week 36: number analyzed (Participants) | 16 | 16
  week 36 | 31.4 (4.0) | 32.3 (5.1)

7. Secondary Outcome: Endosteal Circumference
Description: This was measured at the 20% radius site.
Time Frame: 36 weeks
Population: Sample size reduced due to exclusion of scans with movement artifact and, in later visits, due to attrition as well.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 18 | 20
mm
  Baseline | 16.0 (3.4) | 17.7 (3.6)
  week 18: number analyzed (Participants) | 18 | 16
  week 18 | 17.0 (3.9) | 18.4 (5.1)
  week 36: number analyzed (Participants) | 16 | 16
  week 36 | 16.8 (3.7) | 17.6 (4.0)

8. Secondary Outcome: Polar Section Modulus
Description: This was measured at the 20% radius site.
Time Frame: 36 weeks
Population: Sample size reduced due to exclusion of scans with movement artifact and, in later visits, due to attrition as well.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Calcium+VitD | Placebo
Number analyzed (Participants) | 18 | 20
mm^3
  Baseline | 123.8 (53.6) | 156.2 (76.6)
  week 18: number analyzed (Participants) | 18 | 16
  week 18 | 134.5 (55.1) | 156.8 (91.9)
  week 36: number analyzed (Participants) | 16 | 16
  week 36 | 137.2 (49.2) | 151.9 (75.6)

ADVERSE EVENTS:
Time Frame: Data collected during 36 weeks.
Arm/Group | Calcium+VitD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 11/23 | 8/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium+VitD (N=23) | Placebo (N=24)
Stomach ache (Gastrointestinal disorders) | 5 (5) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3)
Urinary calcium/Creatinine Ratio (Renal and urinary disorders) | 1 (1) | 1 (1)
Increased energy (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Failure to enroll vitamin D deficient patients. The supplements dose were modest. The sample size was small. We may have included too broad a pubertal stage. We did not supplement other micronutrients. We did not include females.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No